CLINICAL TRIAL: NCT00954564
Title: Arthralgia and Medication Adherence in Women With Early Stage Breast Cancer Taking Aromatase Inhibitors: The Breast Cancer Adjuvant Therapy (BCAT) Longitudinal Cohort Study.
Brief Title: Joint Pain and Medication Adherence in Postmenopausal Women Receiving Aromatase Inhibitors
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000650647; UL1RR024975 (NIH); VU-VICC-BRE-0939 (Other: Vanderbilt Ingram Cancer Center); 119475-MRSG-10-169-01-PCSM (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Arthralgia; Breast Cancer
Keywords: arthralgia; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Arthralgia; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: aromatase inhibition therapy - OBSERVATIONAL ONLY — Observational only - as prescribed
Other: medical chart review — Observational only
Other: questionnaire administration — Observational only
Procedure: assessment of therapy complications — Observational only

SUMMARY:
RATIONALE: Gathering information over time about joint pain and stiffness from postmenopausal women with early-stage breast cancer who are receiving aromatase inhibitors may help doctors plan treatment and help patients live more comfortably.

PURPOSE: This observational epidemiologic cohort is designed to study arthralgia, patient-reported outcomes, and medication adherence in postmenopausal women with early-stage breast cancer who are receiving aromatase inhibitors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the incidence, time to onset, prevalence, and clinical and demographic predictors of arthralgia in post-menopausal women with early-stage breast cancer receiving aromatase inhibitors (AI).
* Chart the trajectory of arthralgia symptom severity over the course of AI treatment in these patients.

Secondary

* Measure the impact of arthralgia on sleep quality, depression, and physical function in these patients.
* Develop a roster of current physician-advised or prescribed treatments, including self-management techniques being used for AI-induced arthralgia, for intervention development.

OUTLINE: Patients complete questionnaires about joint pain and stiffness, sleep, depression, physical function, medications and treatment, exercise and social support, demographics, comorbidities, body mass index (BMI), and performance status at baseline and then periodically for approximately 1 year after beginning aromatase inhibitor (AI) therapy.

Patient medical records are reviewed for comorbidities, BMI, use of prior hormone replacement therapy, vitamin D levels and deficiency, performance status, histological stage, prior treatment, and medications at baseline and then periodically for approximately 1 year after beginning AI therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning to begin aromatase inhibitor (AI) therapy or taken fewer than 10 doses of adjuvant AI therapy
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Postmenopausal
* ECOG performance status 0-1
* Able to understand and respond to questions in English
* No condition that would impair the ability to provide informed consent
* No other non-breast cancer condition

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 9 prior doses of AI

Ages: 35 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with breast cancer initiating aromatase inhibitor therapy
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Arthralgia incidence, defined as proportion of the baseline population (those who have taken ≥ 9 doses of aromatase inhibitor [AI]) in which new or worsening joint pain or stiffness is observed at 1, 3, and 12 months after beginning AI therapy | 12 months
Time to onset of arthralgia (continuous variable in weeks) among baseline population | 12 months
Arthralgia point prevalence, defined as proportion of the baseline population with a score of ≥ 2 on any one dimension of the outcome measure at 1, 3, and 12 months after beginning AI therapy | 12 months

SECONDARY OUTCOMES:
Symptom trajectories over the course of treatment | 12 months
Patient well-being: sleep quality, mood, and physical function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liana Castel, PhD, MSPH, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Castel LD, Hartmann KE, Mayer IA, Saville BR, Alvarez J, Boomershine CS, Abramson VG, Chakravarthy AB, Friedman DL, Cella DF. Time course of arthralgia among women initiating aromatase inhibitor therapy and a postmenopausal comparison group in a prospective cohort. Cancer. 2013 Jul 1;119(13):2375-82. doi: 10.1002/cncr.28016. Epub 2013 Apr 10. PMID 23575918